CLINICAL TRIAL: NCT02859454
Title: A Phase II Study of Avelumab in Subjects With Recurrent Respiratory Papillomatosis
Brief Title: Avelumab for People With Recurrent Respiratory Papillomatosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Scott Norberg, D.O., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 160160; 16-C-0160
Record Dates: First submitted 2016-08-06; First posted 2016-08-09 (Estimated); Results first posted 2019-05-14 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-11

CONDITIONS: Recurrent Respiratory Papillomatosis; Juvenile Laryngeal Papilloma; Laryngeal Papilloma, Recurrent; Respiratory Papillomatosis; Human Papilloma Virus
Keywords: PD-L1 Expression; Human Papilloma Virus (HPV); Juvenile-onset Disease; Papillomatous Lesions; Monoclonal Antibody
MeSH Terms: conditions — Recurrent respiratory papillomatosis | interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Avelumab (Experimental): Avelumab 10 mg/kg intravenous (IV) every 2 weeks for up to 6 doses.
  Interventions: Drug: Avelumab

INTERVENTIONS:
Drug: Avelumab — Avelumab 10 mg/kg intravenous (IV) every 2 weeks for up to 6 doses.
  Other Names: Bavencio

SUMMARY:
Background:

Recurrent respiratory papillomatosis (RRP) is a rare disease caused by human papillomavirus. It can cause voice changes, airway compromise, pulmonary lesions, and cancers. Programmed death-ligand 1 (PD-L1) is a protein on cells. It may be able to stop or decrease the immune system s response to viruses such as human papillomavirus. The drug Avelumab interferes with the activity of PD-L1. Researchers want to see if Avelumab treats RRP and study its side effects.

Objective:

To see if Avelumab works in treating RRP and is safe.

Eligibility:

People ages 18 and older with aggressive RRP that has not responded to available treatments

Design:

Participants will be screened with:

Medical history

Previously collected tumor tissue

Physical exam

Blood, urine, and heart tests

Endoscopy procedure: A small tube with a camera is used to look in the nose, throat, larynx, and upper windpipe.

Before starting treatment, participants will have:

Endoscopy under anesthesia. A sample of papilloma will be taken.

Voice handicap questionnaire

Computed tomography (CT) scans

Apheresis: An intravenous (IV) is inserted into an arm vein. White blood cells are separated from the rest of the blood and stored for research. The rest of the blood is returned through the same IV or one in the other arm.

Participants will get the study drug by IV every 2 weeks for up to 12 weeks.

Participants will repeat the previous tests throughout the study.

If they respond to treatment, participants will be evaluated every 6 weeks (3 times), then every 12 weeks (3 times), then every 26 weeks (2 times) until their disease progresses.

Participants will be evaluated 30 days after their last infusion. They will then be contacted annually.

DETAILED DESCRIPTION:
Background

* Recurrent respiratory papillomatosis (RRP) is a rare papillomatous disease of the aerodigestive tract that is caused by the Human Papilloma Virus (HPV).
* RRP can progress to cause airway compromise, fatal pulmonary lesions, and invasive cancers.
* There is no effective systemic therapy for RRP. Patients require repeated interventional procedures for disease control.
* Study of a small number of RRP samples has shown programmed death-ligand 1 (PD-L1) expression by inflammatory mononuclear cells and by papilloma epithelial cells.
* This clinical trial will evaluate the activity of a PD-L1-targeted drug, avelumab, in the treatment of RRP. This drug was selected for its demonstrated activity in a variety of cancers and for its acceptable safety profile.

Objective

-Determine the complete response rate for avelumab in the treatment of patients with RRP.

Eligibility

* Histologically confirmed diagnosis of RRP.
* One of the following:

  * A Derkay anatomic score of 10 or greater and a history of two or more endoscopic interventions in the last 12 months for control of RRP.
  * Pulmonary RRP with pulmonary disease that is measurable by computed tomography scan.
  * Tracheal involvement with RRP that has required either two or more endoscopic interventions in the last 12 months or a tracheostomy.
* Age 18 years or greater.
* Eastern Oncology Cooperative Group Performance Score of 0 or 1.

Design

* Phase II clinical trial
* Simon optimal two-stage design with initial enrollment of 12 patients and expansion to 37 patients if one or more complete response(s) is/are observed in the initial patients.

ELIGIBILITY:
* INCLUSION CRITERIA:

Recurrent Respiratory Papillomatosis (RRP) CRITERIA:

* Histological diagnosis of RRP confirmed by pathology report from a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory.

  -One of the following:
* A Derkay anatomic score of 10 or greater and a history of two or more endoscopic interventions in the last 12 months for control of RRP.
* Pulmonary RRP with pulmonary disease that is measurable by computed tomography scan.
* Tracheal involvement with RRP that has required either two or more endoscopic interventions in the last 12 months or a tracheostomy.

  * Greater than or equal to 18 years of age.
  * Able to understand and sign the Informed Consent Document.
  * Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 or 1.
  * Willing to undergo endoscopic evaluation with biopsies in compliance with this protocol.
  * No systemic therapy for RRP for four weeks prior to treatment.
  * Screening laboratory values must meet the following criteria and should be obtained within 14 days prior to first dose:
* White blood cells (WBC) > 2000/microL
* Neutrophils > 1500/microL
* Platelets > 100 times10(3)/microL
* Hemoglobin > 9.0 g/dL
* Serum creatinine < 1.5 times upper limit of normal (ULN) or creatinine clearance (CrCl) > 30 mL/min (measured or calculated using the Cockcroft-Gault formula below):

  * Female CrCl: (140 - age in years) times weight in kg x 0.85/72 times serum creatinine in mg/dL
  * Male CrCl: (140 - age in years) times weight in kg x 1.00/72 times serum creatinine in mg/Dl
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) less than or equal to 2.5 times ULN; for subjects with documented metastatic disease to theliver, AST and ALT levels less than or equal to 5 times ULN
* Total Bilirubin less than or equal to 1.5 times ULN

  * Sexually active subjects (men and women) and all subjects of reproductive potential must agree to use two methods of contraception: one highly effective and one other effective method for at least 28 days prior, throughout the avelumab treatment and for at least 60 days after avelumab treatment. Highly Effective Methods are defined as: Intrauterine device (IUD), hormonal (birth control pills, injections, implants), tubal ligation and partners vasectomy; Other Effective Methods are defined as: latex condom, diaphragm and cervical cap.
  * Seronegative for human immunodeficiency virus (HIV) antibody. The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune function and thus are likely less responsive to the experimental treatment.
  * Seronegative for hepatitis B antigen, positive hepatitis B tests can be further evaluated by confirmatory tests (Hep B deoxyribonucleic acid (DNA) Quantification (Quant), HBV Viral Load), and if confirmatory tests are negative, the patient can be enrolled.
  * Seronegative for hepatitis C antibody unless antigen negative. If hepatitis C antibody test is positive, then patients must be tested for the presence of antigen by Hep C RNA Quant, Hepatitis C Virus (HCV) Viral Load and be HCV ribonucleic acid (RNA) negative.

EXCLUSION CRITERIA:

* Any severe acute or chronic medical or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; liver, lung disease (with the exception of what is specified in inclusion criteria above), or laboratory abnormalities that, in the opinion of the investigators, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results and in the judgment of the investigator, would make the patient inappropriate for entry into this study. Patients with mild to moderate asthma or chronic obstructive pulmonary disease (COPD) well controlled with oral or inhaled medications are permitted to enroll.
* Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, or psoriasis not requiring systemic treatment, are permitted to enroll.
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled, topical intranasal or intro-ocular steroids, and adrenal replacement doses <10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Prior organ transplantation, including allogeneic stem cell transplantation.
* Prior treatment with an anti-programmed death-ligand 1 (PD-1), anti-PD-L1, anti-programmed death-ligand 2 (PD-L2), anti-cytotoxic T-lymphocyte associated protein 4 (CTLA-4) antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways.
* Patients who are receiving any other investigational agents
* Pregnant or breast feeding. Women of childbearing potential must have a negative pregnancy test at screening. Women of childbearing potential include women who have experienced menarche and who have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or are not postmenopausal. Post-menopause is defined as amenorrhea greater than or equal to 12 consecutive months. Note: women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, anti-estrogens, ovarian suppression or any other reversible reason.
* History of allergy to study drug components.

History of severe hypersensitivity reaction to any monoclonal antibody (Grade greater than or equal to 3 National Cancer Institute (NCI)-Common Terminology Criteria in Adverse Events (CTCAE) v 4.03), any history of anaphylaxis, or uncontrolled asthma (that is, 3 or more features of partially controlled asthma).

* Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (greater than or equal to New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
* Persisting toxicity related to prior therapy of Grade >1 NCI-CTCAE v 4.03; however, alopecia, sensory neuropathy Grade less than or equal to 2 or other Grade less than or equal to 2 adverse events (AEs) not constituting a safety risk based on investigator's judgment are acceptable.
* Known alcohol or drug abuse.
* Vaccination within 4 weeks of the first dose of avelumab and while on trial is prohibited except for administration of inactivated vaccines.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2016-08-06 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2021-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Norberg, DO, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Robbins Y, Friedman J, Clavijo PE, Sievers C, Bai K, Donahue RN, Schlom J, Sinkoe A, Hinrichs CS, Allen C, Abdul Sater H, Gulley JL, Norberg S. Dual PD-L1 and TGF-b blockade in patients with recurrent respiratory papillomatosis. J Immunother Cancer. 2021 Aug;9(8):e003113. doi: 10.1136/jitc-2021-003113. PMID 34462327
- [Derived] Allen CT, Lee S, Norberg SM, Kovalovsky D, Ye H, Clavijo PE, Hu-Lieskovan S, Schlegel R, Schlom J, Strauss J, Gulley JL, Trepel J, Hinrichs CS. Safety and clinical activity of PD-L1 blockade in patients with aggressive recurrent respiratory papillomatosis. J Immunother Cancer. 2019 May 3;7(1):119. doi: 10.1186/s40425-019-0603-3. PMID 31053174
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-C-0160.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Avelumab
Started | 13
Completed | 12
Not Completed | 1
Not completed — PI discretion/off study prior to trtmt | 1

BASELINE CHARACTERISTICS:
Arm/Group | Avelumab
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.95 (15.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13
Patients Who Had Repeated Endoscopic Debulking to Remove Paillomatosis Lesions Prior to Treatment [Count of Participants; unit: Participants] — All patients underwent multiple surgeries as part of standard of care treatment for Recurrent Respiratory Papillomatosis (RRP) prior to enrolling in this protocol.
  Participants | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Laryngotracheal Recurrent Respiratory Papillomatosis (RPP) Who Achieve a Complete Response With Avelumab as Measured by Derkay Score Calculated From Clinical Endoscopy
Description: The Derkay is an objective score based on the number of sites and bulkiness of papillomas within the pharynx, larynx and trachea and a subjective score determined by voice and treating symptoms. Complete response is assessed by The Derkay Staging System which is defined as a physical exam and/or clinic-based flexible nasopharyngolaryngoscopy and/or tracheoscopy, exam under anesthesia with endoscopy and biopsies; no evidence of papillomas on physical exam and/or clinic based flexible nasopharyngolaryngoscopy and/or tracheoscopy; and no evidence of papillomas by exam under anesthesia (sedation or general anesthesia) with endoscopy and biopsies.
Time Frame: Disease response was performed at 6 and 12 weeks after the first dose of Avelumab. Patients who experience a complete response will be evaluated every 6 weeks x 3, then every 12 weeks x 3, then every 26 weeks x 2 or until disease progression,up to 3 years
Population: Nine of twelve patients had evaluable laryngotracheal disease as assessed by clinical endoscopy.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab
Number analyzed (Participants) | 9
Participants | 0

2. Primary Outcome: Number of Patients With Pulmonary Recurrent Respiratory Papillomatosis (RPP) Who Achieve a Complete Response With Avelumab as Measured by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 Calculated From Chest Computed Tomography (CT) Scans
Description: Complete response is measured by The Response Criteria in Solid Tumors (RECIST) v1.1 calculated from chest CT scans. Complete response is absence of disease (e.g., lesions) by imaging.
Time Frame: as for outcome 1
Population: Four of twelve patients had evaluable pulmonary disease as assessed by CT scan.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab
Number analyzed (Participants) | 4
Participants | 0

3. Secondary Outcome: Effect of Treatment With Avelumab on Voice Handicap Index-10 Score
Description: The Voice Handicap Index-10 questionnaire (as measured by derkay score) consists of 10 questions and determines whether a participant has a voice handicap. The scoring options for each question range from 0 (for never) to 4 (for always). The total scores (combined value from all 10 questions) range from 0 - 40. Higher scores represent a worse voice handicap. Lower scores represent a less voice handicap.
Time Frame: Baseline, 6 weeks, and 12 weeks after the first dose of Avelumab.
Population: Only one participant in each row contributed data in each row.
Measure: Number; unit: scores on a scale
Groups:
- All Participants at Baseline: All participants Voice Handicap Index-10 Score at Baseline.
  Avelumab 10 mg/kg intravenous (IV) every 2 weeks for up to 6 doses. Avelumab: Avelumab 10 mg/kg intravenous (IV) every 2 weeks for up to 6 doses.
- All Participants at 6 Weeks: All participants Voice Handicap Index-10 Score at 6 Weeks.
  Avelumab 10 mg/kg intravenous (IV) every 2 weeks for up to 6 doses.
  Avelumab: Avelumab 10 mg/kg intravenous (IV) every 2 weeks for up to 6 doses.
- All Participants at 12 Weeks: All participants Voice Handicap Index-10 Score at 12 Weeks.
  Avelumab 10 mg/kg intravenous (IV) every 2 weeks for up to 6 doses.
  Avelumab: Avelumab 10 mg/kg intravenous (IV) every 2 weeks for up to 6 doses.
Arm/Group | All Participants at Baseline | All Participants at 6 Weeks | All Participants at 12 Weeks
Number analyzed (Participants) | 12 | 12 | 12
scores on a scale
  Patient 1: number analyzed (Participants) | 1 | 1 | 1
  Patient 1 | 26 | 22 | 23
  Patient 2: number analyzed (Participants) | 1 | 1 | 1
  Patient 2 | 9 | 12 | 3
  Patient 3: number analyzed (Participants) | 1 | 1 | 1
  Patient 3 | 40 | 37 | 38
  Patient 4: number analyzed (Participants) | 1 | 1 | 1
  Patient 4 | 17 | 16 | 16
  Patient 5: number analyzed (Participants) | 1 | 1 | 1
  Patient 5 | 12 | 2 | 1
  Patient 6: number analyzed (Participants) | 1 | 1 | 1
  Patient 6 | 19 | 0 | 0
  Patient 7: number analyzed (Participants) | 1 | 1 | 1
  Patient 7 | 40 | 21 | 18
  Patient 8: number analyzed (Participants) | 1 | 1 | 1
  Patient 8 | 30 | 35 | 29
  Patient 9: number analyzed (Participants) | 1 | 1 | 1
  Patient 9 | 37 | 40 | 40
  Patient 10: number analyzed (Participants) | 1 | 1 | 1
  Patient 10 | 18 | 11 | 12
  Patient 11: number analyzed (Participants) | 1 | 1 | 1
  Patient 11 | 18 | 9 | 0
  Patient 13: number analyzed (Participants) | 1 | 1 | 1
  Patient 13 | 18 | 19 | 15

4. Secondary Outcome: Number of Patients With Laryngotracheal Recurrent Respiratory Papillomatosis (RPP) Who Achieve a Partial Response With Avelumab as Measured by Derkay Score Calculated From Clinical Endoscopy
Description: Partial response is assessed by flexible nasopharyngolaryngoscopy and/or tracheoscopy using the Derkay staging system if the patient does not have pulmonary disease. The Derkay is an objective score based on the number of sites and bulkiness of papillomas within the pharynx, larynx and trachea and a subjective score determined by voice and treating symptoms. Partial response is a decrease in Derkay anatomic score of 30% or greater.
Time Frame: as for outcome 1
Population: Nine of twelve patients had evaluable laryngotracheal disease as assessed by clinical endoscopy.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab
Number analyzed (Participants) | 9
Participants | 6

5. Secondary Outcome: Number of Patients With Pulmonary Recurrent Respiratory Papillomatosis (RPP) Who Achieve a Partial Response With Avelumab as Measured by the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 Calculated From Chest Computed Tomography (CT) Scans
Description: Partial response assessed by imaging using RECIST v1.1. is defined as a ≥ 30% decrease in the sum of the longest diameters of target lesions compared with baseline.
Time Frame: Disease response was performed at 6 and 12 weeks after the first dose of Avelumab. Patients who experience a complete response will be evaluated every 6 weeks x 3, then every 12 weeks x 3, then every 26 weeks x 2 or until disease progression, up to 3 year
Population: Four of twelve patients had evaluable pulmonary disease as assessed by CT scan.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab
Number analyzed (Participants) | 4
Participants | 0

6. Secondary Outcome: Duration of Clinical Responses to Avelumab
Description: The duration of clinical responses to Avelumab is calculated from the protocol end of treatment endoscopic debulking to the next clinically indicated endoscopic debulking procedure.
Time Frame: Disease response was performed at 6 and 12 weeks after the first dose of Avelumab. Patients who experience a complete response will be evaluated every 6 weeks x 3, then every 12 weeks x 3, then every 26 weeks x 2 or until disease progression,up to 4.5 yrs
Population: 5/12 participants were evaluable for this outcome measure.
Measure: Mean (Full Range); unit: Months
Arm/Group | Avelumab
Number analyzed (Participants) | 5
Months | 14.7 [4.5 to 51]

7. Secondary Outcome: Number of Participants With Serious and Non-serious Adverse Events
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Common Terminology Criteria in Adverse Events (CTCAE v4.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 28 months and 20 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab
Number analyzed (Participants) | 13
Participants | 13

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 28 months and 20 days.
Arm/Group | Avelumab
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 2/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avelumab (N=13)
Cardiac disorders - Other, Stress cardiomyopathy (Cardiac disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avelumab (N=13)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (3)
Anxiety (Psychiatric disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cardiac disorders - Other, Stress cardiomyopathy (Cardiac disorders) | 1 (1)
Cardiac troponin I increased (Cardiac disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 5 (9)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2)
Dysgeusia (Nervous system disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Ejection fraction decreased (Cardiac disorders) | 1 (2)
Fatigue (General disorders) | 7 (11)
Fever (General disorders) | 3 (4)
Headache (Nervous system disorders) | 4 (7)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 8 (41)
Hyperthyroidism (Endocrine disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (3)
Hypotension (Vascular disorders) | 1 (1)
Infections and infestations - Other, yeast infection (Infections and infestations) | 1 (1)
Infusion related reaction (General disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 2 (2)
Malaise (General disorders) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (8)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (2)
Pain (General disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3)
Sinus bradycardia (Cardiac disorders) | 5 (10)
Sinus tachycardia (Cardiac disorders) | 3 (8)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (3)
White blood cell decreased (Investigations) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/54/NCT02859454/Prot_SAP_002.pdf
  • Informed Consent Form (2020-12-30): https://cdn.clinicaltrials.gov/large-docs/54/NCT02859454/ICF_003.pdf